CLINICAL TRIAL: NCT03818802
Title: A Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Effects of Vitamin B3 Derivative Nicotinamide Riboside (NR) in Bone, Skeletal Muscle and Metabolic Functions in Aging
Brief Title: Effects of Vitamin B3 Derivative Nicotinamide Riboside (NR) in Bone, Skeletal Muscle and Metabolic Functions in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eduardo N. Chini, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-000224
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-04

CONDITIONS: Healthy Elderly Volunteers
Keywords: NAD boosting therapy; Nicotinamide Riboside; NAD precursors; Aging
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 48 subjects (24 placebo vs. 24 NR) considering a dropout rate of 20%. Patients will be screened at outpatient clinic visit by the research team before the enrollment. For those subjects interested and qualified it will be offered participation in this trial. Once consent has been obtained baseline values will be established and subjects will begin treatment and followed for 4.5 months. After 4.5 months, a structured exercise regimen will be implemented in addition to the NR/placebo treatment and the patients will be followed for 6 weeks more, completing 6 months.
Who Masked: Participant, Investigator
Masking Description: This protocol will employ a blinded design so that the participant, study personnel, and investigators will not know subject group assignment status. The unblinding would be done by contacting the research pharmacy. While the safety of the subject always comes first, it is still important to seriously consider if unmasking/unblinding the study therapy is necessary to ensure a subject's safety. The unmasking/unblinding will happen only when there is a serious adverse event; in this case this event will be logged in the specific Case Report Form for Serious Adverse Event (SAE) that is part of this protocol. However, in cases where unmasking/unblinding was not associated with an SAE, such actions will be reported in a same timeline requirements for reporting of SAEs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide Riboside (Active Comparator): NR is a single chemical moiety containing nicotinamide and ribose. The investigational product is a synthetic NR that is nature-identical to naturally-occurring NR, does not induce flushing or pruritus and has no effect on lipid levels.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Correspondent placebo, a pill not containing the active component.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — It will be administered a total of 1000 mg/day of NR in a regimen of 500mg every 12 hours by mouth for 4.5 months. After 4.5 months, an advanced individual training (AIT) will be implemented in addition to administration of 1000mg/day (500mg every 12 hours) for 6 weeks more, completing total of 6 months.
  Arms: Nicotinamide Riboside
Dietary Supplement: Placebo — It will be administered a correspondent placebo with the same shape and color as the active pill 12 hours by mouth for 4.5 months. After 4.5 months, an advanced individual training (AIT) will be implemented in addition to administration of correspondent placebo every 12 hours for 6 weeks more, completing total of 6 months.
  Arms: Placebo

SUMMARY:
Researchers are trying to determine if the vitamin B3 derivative Nicotinamide Riboside (NR) has any effects in bone, skeletal muscle, and metabolic functions and structure in aging.

DETAILED DESCRIPTION:
Primary Objective: To assess the effect of "NAD boosting" through NR intake in skeletal muscle and bone metabolism function, and biochemical evidence of improvement of DNA damage repair in healthy elderly female patients with and without exercise.

Secondary Objective: To assess the effect of NR in metabolic functions of glucose and lipid profile as well as to determine the safety of long term administration of NR in healthy elderly female patients with and without exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly female subjects between 65 and 80 years of age

Exclusion Criteria:

* General Exclusion Criteria

  * Subjects who participate in regular structured exercise more than 2 hours and 30 min per week or 1hour and 15 min of vigorous exercise per week.
  * Unwilling to comply with the follow-up schedule
  * Inability or refusal to give informed consent by the patient
  * Subject who takes multivitamins containing vitamin B3 derivatives in a dose > 200 mg/day
  * Participation in another investigational drug study within 1 year of treatment
* Laboratory Exclusion Criteria

  * Serum 25-hydroxyvitamin D < 15 ng/ml
  * Serum phosphorus > 5 mg/dL
  * Serum alkaline phosphatase 50% above normal limit
  * Serum aspartate transaminase 50% above normal limit
  * Serum calcium > 10.5 mg/dL
  * Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min Creatinine Clearance < 50%
  * Poorly controlled Diabetes Mellitus (HbA1c>8)
* Clinical History Exclusion Criteria

  * Confirmed diagnosis of Diabetes Mellitus in use of insulin
  * Subjects presenting systolic BP>180 mmHg or a diastolic BP>90 mmHg on initial evaluation
  * Previous diagnosis of liver disease
  * Previous chronic kidney disease stages III and IV
  * Malignancy
  * Malabsorption syndrome
  * Hypo- or Hyperparathyroidism
  * Acromegaly
  * Cushing's syndrome
  * Hypopituitarism
  * Severe chronic obstructive pulmonary disease
  * Congestive heart failure
  * Musculoskeletal disorder
  * History of rheumatoid arthritis
  * Previous gastric bypass surgery
  * Clinical history of osteoporotic fracture (spine, hip, or distal forearm) within past year
  * Extreme of BMI (≤ 18.5 kg/m2 or ≥ 40 kg/m2)
* Medication Exclusion Criteria

  * History of methotrexate therapy
  * History of denosumab therapy
  * History of oral or inhaled corticosteroid use > 3 months
  * Current use of anticoagulants in general
  * Anticonvulsant therapy (within previous year)
  * Sodium fluoride (any history)
  * Treatment within the past 3 years with bisphosphonates
  * Treatment within the past 3 years with parathyroid hormone
  * Treatment within the past 3 years with calcitonin
  * Treatment within the past 3 years with estrogen
  * Treatment within the past 3 years with selective estrogen receptor modulator

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2 max) test | 6 months
  Maximal oxygen uptake (VO2 max) test measures the maximum rate of oxygen consumption during incremental exercise (exercise of increasing intensity) and reflects the cardiorespiratory fitness of an individual and is an important determinant of their endurance capacity during prolonged exercise.
Skeletal muscle function | 6 months
  The 6-minute walk test (6MWT) quantifies the distance a person can walk in six minutes and will be used to document the mobility/functional status of a patient. Originally developed to evaluate the physical capacity of patients with cardiopulmonary diseases, the test has been used to assess treatment effects, physical function status, and to predict morbidity and mortality in several patient populations including frail older adults.
Short Physical Performance Battery (SPPB) | 6 months
  The SPPB captures domains of strength, endurance, and balance and is highly predictive of subsequent disability.
Respiration rate on muscle biopsy samples | 6 months
  The samples will be analyzed for respiration rate in isolated mitochondria and permeabilized fibers
PCR on muscle biopsy samples | 6 months
  RT-PCR for gene expression
Immunoblot on muscle biopsy samples | 6 months
  Immunoblot in skeletal lysates for protein expression
Bone metabolism | 6 months
  Serum Carboxy-terminal Telopeptide (CTX), tartrate-resistant acid phosphatase isoform type 5b (TRAP5b), Amino-terminal Pro-peptide (P1NP), and osteocalcin will all be measured to monitor bone turnover markers.

SECONDARY OUTCOMES:
Glucose profile | 6 months
  Serum glucose measure
Insulin | 6 months
  Serum insulin measure
Lipid profile | 6 months
  Blood cholesterol measure
Hemoglobin A1C | 6 months
  Hb A1C measure in blood sample
Oral glucose tolerance test | 6 months
  An 18-gauge cannula will be inserted in a retrograde fashion into a dorsal hand vein of the non-dominant arm. The hand will be placed in a heated box (55°C) to enable sampling of arterialized venous blood. Blood will be drawn at 0 (baseline), 10, 20, 30, 60, 90, and 120 minutes for the measurement of glucose, insulin, and C-peptide concentrations. After the baseline blood draw, subjects will ingest 75 g of glucose over a period of 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo N Chini, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials